CLINICAL TRIAL: NCT06581952
Title: Chinese Poem Writing for Improving Mental Wellbeing of Adult Volunteers Serving for People Recovering From Mental Illness
Brief Title: Chinese Poem Writing for Improving Mental Wellbeing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Metropolitan University (Other)
Collaborators: Bestreben Drama Association Limited (Unknown)
Responsible Party: Principal Investigator, Dr Agnes LAI Yuen Kwan, Associate Professor, Hong Kong Metropolitan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: HE-SF2024/19
Record Dates: First submitted 2024-06-13; First posted 2024-09-03 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Well-Being, Psychological; Happiness
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Two poem writing sessions (Experimental): The intervention consists of two sessions of poem writing. Each session lasts for 3 hours. The instructors for each session will include two experienced Chinese teachers or drama directors from Bestreben Drama Association Limited. Adherence to the protocol will be evaluated by two independent reviewers.
  Interventions: Behavioral: Poem writing

INTERVENTIONS:
Behavioral: Poem writing — The poem themes will focus on accomplishment moments, joyful moments, and gratitude. Participants will be motivated to write at least one poem in each session. The instructor will lead the participants to improve the poem after the participants complete the first draft. The participants will be encouraged to perform in reading their completed poem, sharing their feelings and expressing the meaning of the poems during the session.
  In the second session, participants will be invited to do a poem reading performance using one of their newly written poems.

SUMMARY:
This research proposal aims to explore the impact of poem writing on the well-being of adult volunteers serving patients recovering from mental illness in Hong Kong. The research design was a single-arm intervention study with 30 participants. The intervention consists of two sessions of poem writing, each lasting for 3 hours, led by experienced Chinese teachers or drama directors. The themes of the poems will focus on accomplishment, joy, and gratitude. The primary outcomes are mental well-being and happiness, measured using the Short Warwick-Edinburgh Mental Well-being Scale and a single-item happiness scale. Feasibility outcomes include recruitment rate, retention rate, and acceptability of the interventions. Secondary outcomes include depressive symptoms, anxiety, interest in poem writing, perceived benefits after the activity, and the number of successfully written poems. The proposal also includes plans for in-depth interviews with participants to gather qualitative data. The results will be analyzed descriptively and narratively, with no efficacy statistical tests due to the nature of this feasibility study. The proposal highlights the potential of poem writing as a therapeutic tool for volunteers serving patients recovering from mental illness, enhancing their overall well-being.

DETAILED DESCRIPTION:
This research proposal aims to explore the impact of poem writing on the well-being of adult volunteers serving patients recovering from mental illness in Hong Kong.The research design was a single-arm intervention study with 30 participants. The intervention consists of two sessions of poem writing, each lasting for 3 hours, led by experienced Chinese teachers or drama directors. The themes of the poems will focus on accomplishment, joy, and gratitude.

The primary outcomes are mental well-being and happiness, measured using the Short Warwick-Edinburgh Mental Well-being Scale and a single-item happiness scale. Feasibility outcomes include recruitment rate, retention rate, and acceptability of the interventions. Secondary outcomes include depressive symptoms, anxiety, interest in poem writing, perceived benefits after the activity, and the number of successfully written poems.

Moreover, the proposal includes plans for in-depth interviews with participants to gather qualitative data. The results will be analyzed descriptively and narratively, with no efficacy statistical tests due to the nature of this feasibility study.

Apart from that, the process evaluation will be done by the instructors after the end of the second class, including the teachers, speakers and the leaders of each group. This act aims to evaluate the effectiveness of using the app in creating and writing poems, as well as the feelings after class on the instructors. An evaluation analysis will be made after the collection of data.

The proposal underscores the potential of poem writing as a therapeutic tool for volunteers serving patients recovering from mental illness, enhancing their overall well-being. Poem writing not only allows volunteers to express their thoughts, emotions, and experiences, but also enhances their self-esteem by validating their feelings and providing a sense of accomplishment. Volunteers working with individuals recovering from mental illness often encounter intense emotions. Writing poems allows them to channel these emotions constructively, preventing burnout and fostering resilience. Furthermore, the act of creating poems can be joyful and fulfilling. Volunteers experience a sense of flow, where time seems to disappear as they immerse themselves in the creative process. Lastly, incorporating poem writing into volunteer programs can be a powerful tool for enhancing both the volunteers' and the patients' well-being, self-esteem, and emotional resilience. Volunteers can find solace, connection, and purpose through their poetic expressions, ultimately benefiting both themselves and the individuals they serve.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers serving for people recovering from mental illness or other community residents
* Aged 18 years old and above
* Able to understand Cantonese and read Chinese

Exclusion Criteria:

* Physically or mentally unable to communicate
* Unwilling to participate or give consent
* Being involved in other similar activities or research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in well-being | Baseline, 2 weeks, 4 weeks, 12 weeks
  The 7-item Short Warwick-Edinburgh Mental Well-being Scale with the 5-point Likert scale ("1" means "None of the time", while "5" means "All the time") will be used to measure participants' well-being. The score is calculated by summing up all seven items and with a range of 7 to 35. A higher score indicates a higher positive mental well-being.
Changes in happiness | Baseline, 2 weeks, 4 weeks, 12 weeks
  Happiness of participants across four timeslots were measured by a single item question, which was "How happy do you think you are" (from "0" = "Not at all" to "10" = "very happy").

SECONDARY OUTCOMES:
Changes in depressive symptoms | Baseline, 2 weeks, 4 weeks, 12 weeks
  The Patient Health Questionnaire (PHQ)-9 will be used to measure depressive symptoms among all participants. Participants rate the frequency of nine symptoms over the past two weeks on a 4-point Likert scale (from "0" = "Not at all" to "3" = "Nearly every day"). The total score ranges from 0 to 27, with higher scores indicating a greater severity of depressive symptoms.
Changes in perceived knowledge about limericks (Chinese poem) | Baseline, 2 weeks, 4 weeks, 12 weeks
  The changes in participants' perceived knowledge about limericks (Chinese poem) were measured by a single item question, which was "How much do you know about limericks", scoring from "0" (very little understanding) to "10" (very much understanding).
Changes in perceived interest in limericks writing | Baseline, 2 weeks, 4 weeks, 12 weeks
  The changes in participants' perceived interest in limericks writing were measured by a single item question, which was "How interested are you in limerick writing?", scoring from "0" (very little interest) to "10" (very much interest).
Changes in perceived confidence in limericks writing | Baseline, 2 weeks, 4 weeks, 12 weeks
  The changes in participants' perceived confidence in limericks writing were measured by a single item question, which was "How confident are you in writing limerick?", scoring from "0" (very little confidence) to "10" (very much confidence).
Changes in perceived usefulness of limericks writing | Baseline, 2 weeks, 4 weeks, 12 weeks
  The changes in participants' perceived usefulness of limericks writing were measured by three aspects, which were "improving happiness", "improving accomplishment" and "developing new hobbies", all of them were scoring from "0 " (very little help) to "10" (very much help).
The number of successfully written poems | 2 weeks, 4 weeks, 12 weeks
  The actual number of successfully written poems will be reported subjectively by participants.

OTHER OUTCOMES:
Recruitment rate | 12 weeks
  The percentage of enrolled participants in the approached participants
Retention rate | 2 weeks, 4 weeks
  The percentage of adhered participants in the enrolled participants
Acceptability of the intervention | 2 weeks, 4 weeks
  Participants' engagement level (from 0 "did not engage at all" to 10 "totally engaged") and happiness level (from 0 "not at all" to 10 "very happy") after joining the activity, satisfaction towards the activity (from 0 "not at all" to 10 "very satisfied"), willingness to write poems after the activity (from 0 "not at all" to 10 "very willing to") and willingness to attend similar activities in the future (from 0 "not at all" to 10 "very willing to"). An average score will be calculated.

CONTACTS AND LOCATIONS:
Locations (1):
- Jockey Club Institute of Healthcare, Hong Kong Metropolitan University, Hong Kong, Hong Kong